CLINICAL TRIAL: NCT04522622
Title: Treatment of Adynamic Bone Disorder With Parathyroid Hormone in Patients With Chronic Kidney Disease
Brief Title: Treatment of Adynamic Bone Disorder With Parathyroid Hormone in Chronic Kidney Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ditte Hansen (Other)
Collaborators: Odense University Hospital (Other); Steno Diabetes Center Copenhagen (Other); Rigshospitalet, Denmark (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ditte Hansen, MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANDYNAMIC BONE; 2018-003888-56 (EudraCT Number)
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Adynamic Bone Disease; Chronic Kidney Diseases; Cardiac Disease; Chronic Kidney Disease-Mineral and Bone Disorder
Keywords: Fracture risk; Teriparatide
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Diseases; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Teriparatide; X-Rays; Heart Function Tests; Blood Specimen Collection; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriparatide (Experimental): Patients receive teriparatide 20 micrograms once daily for 18 months
  Interventions: Drug: Teriparatide; Diagnostic Test: DXA,VFA, X-ray, HR-pQCT, 18-F NAF PET/CT; Procedure: Bone biopsy; Diagnostic Test: Cardiac tests; Other: Blood and urine samples and physical examination
- Controls (Other): Controls receive no treatment with teriparatide
  Interventions: Diagnostic Test: DXA,VFA, X-ray, HR-pQCT, 18-F NAF PET/CT; Procedure: Bone biopsy; Diagnostic Test: Cardiac tests; Other: Blood and urine samples and physical examination

INTERVENTIONS:
Drug: Teriparatide — 20 micrograms
  Other Names: Terrosa
  Arms: Teriparatide
Diagnostic Test: DXA,VFA, X-ray, HR-pQCT, 18-F NAF PET/CT — All participants undergo DXA and VFA or X-ray scans 3 times during the study. Some participants (those connected to Herlev) are offered 18F NAF PET/CT scans at baseline and after 12 months and some participants (those connected to Odense University Hospital and Aalborg University Hospital) are offered HR-pQCT scans at baseline and after 12 months. The 18F-NAF PET/CT and HR-pQCT are optional, so it is not a must to have these procedures done to participate in the study.
Procedure: Bone biopsy — All participants are invited to undergo a bone biopsy after 12 months, but it is not a must to have the procedure done to participate in the study.
Diagnostic Test: Cardiac tests — All participants are invited to undergo 24-hour blood pressure measurements and pulse wave measurements at baseline and after 18 months, but it is not a must to have these procedures done to participate in the study.
Other: Blood and urine samples and physical examination — All participants must undergo a physical examination and deliver blood and urine samples in order to participate in the study.

SUMMARY:
This study is a 1:1 randomized controlled trial with an intervention for 18 months and a follow up period of 12 months. The purpose of the study is to assess the safety and efficacy of recombinant human parathyroid hormone for treatment of adynamic bone disorder in patients with chronic kidney disease.

DETAILED DESCRIPTION:
This study is a 1:1 randomized controlled trial with an intervention for 18 months and a follow up period of 12 months.

The study will explore if treatment with recombinant human parathyroid hormone (PTH) improves bone turnover and bone mineral density (BMD), and thereby prevents the high risk of fracture in patients with chronic kidney disease (CKD).

Disturbed bone metabolism is related to increased risk of cardiovascular disease in patients with CKD. This study also wishes to examine of treatment with recombinant PTH improves cardiovascular parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CKD stage 4-5D (eGFR ≤29 ml/min) according to Kidney Disease Improving Global Outcomes(KDIGO) definition
* DXA scan with a T-score at the total hip, femoral neck or lumbar spine (L1-4) ≤-2 (or Z-score ≤-2) in a minimum of 2 vertebraes (for patients with active oral prednisolone treatment ≥ 5 mg/day for minimum 3 months the T-score or Z-score limit i < -1) and/or former fragility fracture (vertebral, hip, for- or upper arm, ankle) assessed with VFA or x-ray of the columna
* Patients with expected adynamic bone disorder, based on BSAP≤21 µg/l or biopsy-verified low bone turnover

Exclusion Criteria:

* Hypercalcemia defined as sustained ionized calcium >1.35 mmol/l
* Previous fracture withon the last 6 months *Patients may be rescreened after the 6 months
* Previous calciphylaxis
* Thyroid disturbances not adequately treated based on the opinion by the clinician *Patients may be rescreened after treatment optimization
* Treatment with digoxin
* Paget's disease or other metabolic bone disorders
* Antiresorptive or bone anabolic medication during the last 24 months (for bisphosphonates it is only during the last 12 months)
* Former or present malignant disease (except skin basal or planocellular carcinoma)
* Previous external beam or implant radiation therapy to the skeleton
* Patients who have undergone a kidney transplantation within the last 12 months
* 25 hydroxyvitamin D2 and D3 <50 nmol/l *Patients may be rescreened after correction
* Inability to administer teriparatide
* Reduced liver function *Alanine Aminotransferase (ALAT) >3x upper limit of normal or bilirubin > 2x upper limit of normal
* Pregnancy, lactation or fertile women (post-menopausal females are not considered fertile) not using safe anticonception (the following contraceptive methods are considered appropriate: Intrauterine device (IUD) or hormonal anticontraceptive (oral contraceptives, implant, transdermal patches, vaginal ring or depot injection)).
* Hypersensitivity to the active substance in teriparatide or to any of the excipients or content
* Inability to provide informed consent
* Medical conditions or treatments that may interfere with assessments of the outcomes of the trial
* Drug or alcohol abuse
* Unable to participate in a clinical study based on the judgement by the local investigator
* For those participating in the bone biopsy procedure: 1) Hypersensitivity to any of the tetracyclines or to any of the excipients or content, 2) Treatment with anticoagulants (vitamin K antagonists, Non-vitamin K Antagonist Oral Anticoagulants (NOAC), unfractionated or low-molecular heparin or antiplatelet agents that, due to clinical indication can't be paused, 3) Disturbances in thrombosis and/or haemostasis
* For those participating in pulse wave measurements: 1) Atrial fibrillation, 2) Aorta stenosis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in bone specific alkaline phosphatase (BSAP) | Baseline and 18 months
  The difference between treated and controls in changes from baseline to 18 months in bone specific alkaline phosphatase

SECONDARY OUTCOMES:
Number of patients who no longer has adynamic bone disorder based on a BSAP >21 µg/l | Baseline and 18 months. It is also measured through study completion, an average of 30 months
  Changes between baseline and 18 months as well as differences between treated and controls.
BMD at the lumbar spine, antebrachium, femoral neck and total hip | Baseline and 18 months. The scan is also performed at 30 months
  Changes between baseline and 18 months as well as differences between treated and controls
Incidence of fragility fractures and vertebral fractures assessed using x-ray of columna or vertebral fracture assessment (VFA) | Baseline and 18 months. The scan is also performed at 30 months
  Changes between baseline and 18 months as well as differences between treated and controls
Bone microarchitecture assessed using high-resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline and 12 months
  Changes between baseline and 12 months as well as differences between treated and controls. The HR-pQCT scan is a voluntary procedure.
Volumetric BMD assessed using high-resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline and 12 months
  Changes between baseline and 12 months as well as differences between treated and controls. The HR-pQCT scan is a voluntary procedure.
Bone geometry assessed using high-resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline and 12 months
  Changes between baseline and 12 months as well as differences between treated and controls. The HR-pQCT scan is a voluntary procedure.
Bone strength assessed using high-resolution peripheral quantitative computed tomography (HR-pQCT) | Baseline and 12 months
  Changes between baseline and 12 months as well as differences between treated and controls. The HR-pQCT scan is a voluntary procedure.
Regional bone formation using 18F-Sodium Fluoride Positron Emission Tomography/Computed Tomography (18F-NAF PET/CT) | Baseline and 12 months
  Changes between baseline and 12 months as well as differences between treated and controls. The 18F-NAF PET/CT is a voluntary procedure.
Changes in p-PTH | Baseline and 18 months. Some of them are also measured during follow up.
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in p-phosphate | Baseline and 18 months. Some of them are also measured during follow up.
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in p-magnesium | Baseline and 18 months. Some of them are also measured during follow up.
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in calcium | Baseline and 18 months. Some of them are also measured during follow up.
  P-ionised calcium. Changes between baseline and 18 months as well as differences between treated and controls.
Bone histomorphometry | 12 months
  Static and dynamic bone histomorphometry classified by the bone Turnover Mineralization Volume (TMV) classification assessed by bone biopsy. Performed after 12 months. This is a voluntary procedure.
Changes in Intact Procollagen type 1 N-terminal Propeptide (P1NP) | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in total P1NP | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in Tartrate-Resistant Acid Phosphatase 5b (TRAP5b) | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in sclerostin | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in Receptor Activator of Nuclear factor Kappa-B Ligand (RANKL) | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in Osteoprotegerin (OPG) | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in Fibroblast Growth Factor 23 (FGF-23) | Baseline and 18 months. They are also measured during follow up
  Changes between baseline and 18 months as well as differences between treated and controls.
24-hour blood pressure | Baseline and 18 months
  Changes between baseline and 18 months as well as differences between treated and controls. These are voluntary procedures.
Pulse wave measurements including velocity | Baseline and 18 months
  Changes between baseline and 18 months as well as differences between treated and controls. These are voluntary procedures.
Changes in cardiovascular marker Calciprotein Particles (CPP)/T50 | Baseline and 18 months
  Changes between baseline and 18 months as well as differences between treated and controls.
Changes in cardiovascular marker N-Terminal pro B-type Natriuretic Peptide (NT-proBNP) | Baseline and 18 months
  Changes between baseline and 18 months as well as differences between treated and controls.
Adverse reactions | From baseline to 18 months
  The incidence of adverse reactions in treated patients. This is examined during the entire study.
Bone microstructure | 12 months
  Bone mictrostructure by micro-compyter tomography of the bone biopsy
Bone histology | 12 months
  Detailed histology of underlying cellular mechanisms using a combination of immunostainings and advanced in situ hybridizations on the bone biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, MD, PhD, Principal Investigator — Department of Nephrology, Herlev and Gentofte Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Herlev and Gentofte Hospital, Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
As of now we have no plan to share Individual Participant Data (IPD) with other researchers